CLINICAL TRIAL: NCT05251584
Title: Effects of Topical Gentamicin on the Prevention of Peritoneal Dialysis Related Infection Caused by Pseudomonas Aeruginosa
Brief Title: Effects of Topical Gentamicin on the Prevention of Peritoneal Dialysis Related Infection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Phramongkutklao College of Medicine and Hospital (Other)
Collaborators: Silpakorn University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PDRI-2021
Record Dates: First submitted 2022-01-04; First posted 2022-02-22 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: Peritoneal Dialysis-related Infection
Keywords: Peritoneal dialysis-related infection; Infectious peritonitis; Exit-site infection; Infection rate; Drug susceptibility
MeSH Terms: interventions — Mupirocin; Gentamicins

STUDY DESIGN:
Intervention Model Description: Single group: topical mupirocin ointment retrospective period compare with gentamicin prospective period
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mupirocin and Gentamicin (Experimental): 2% mupirocin ointments apply at exit-site once daily after wound cleaning before recruit in the study then use 0.1% gentamicin cream apply at exit-site once daily after wound cleaning after entry to the study.
  Interventions: Drug: Mupirocin; Drug: Gentamicin

INTERVENTIONS:
Drug: Mupirocin — Apply mupirocin ointments for prevention of peritoneal dialysis-related infection between 1 January 2021 to 31 December 2021
  Other Names: BACIDAL
Drug: Gentamicin — Apply gentamicin creams for prevention of peritoneal dialysis-related infection for 1 year start after 1 January 2022
  Other Names: GENTREX

SUMMARY:
Peritoneal dialysis-related infection is a complication that leads to peritoneal dialysis catheter removal or patient death. The present study aimed to investigate peritoneal dialysis-related infection, causative pathogens resulting in topical 2% mupirocin ointments period compare with 0.1% gentamicin cream period. Rate of catheter removal, time to first peritoneal dialysis-related infection after apply gentamicin cream.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 20 years
* End stage renal disease patients on peritoneal dialysis follow up at Phramongkutklao hospital's peritoneal dialysis clinic between January 1, 2021 to March 31, 2023
* Start peritoneal dialysis or follow up at Phramongkutklao hospital's peritoneal dialysis clinic at least 90 days before recruited
* Use topical mupirocin ointment for prevention of peritoneal dialysis-related infection between January 1, 2021 to December 31, 2021
* Can be used LINE application throughout the study

Exclusion Criteria:

* Allergy to gentamicin or components
* Previous systemic antibiotics use within 90 days before recruited
* Previous peritoneal dialysis-related infection within 28 days before recruited
* Immunosuppressants used
* Prospective follow up less than 2 months
* Don't sign informed consent

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
Rate of Exit-site infection in mupirocin compared with gentamicin group | All exit-site infection episodes occurred last year in mupirocin group and all exit-site infection episodes have occurred after apply 0.1% grntamicin cream for 1 year.
  Exit-site infection diagnosis by physician. Retrospective data collection from patient's medical records in mupirocin group Prospective data collection from patient's medical records in gentamicin group.
Rate of Infectious peritonitis in mupirocin compared with gentamicin group | All infectious peritonitis episodes occurred last year in mupirocin group and all infectious peritonitis episodes have occurred after apply 0.1% grntamicin cream for 1 year.
  Infectious peritonitis diagnosis by physicians. Retrospective data collection from patient's medical records in mupirocin group Prospective data collection from patient's medical records in gentamicin group

SECONDARY OUTCOMES:
Number and percentage Causative pathogens of Exit-site infection in mupirocin compared with gentamicin group | All pathogenic organisms of exit-site infection episodes occurred last year in mupirocin group and all pathogenic organisms of exit-site infection episodes have occurred after apply 0.1% grntamicin cream for 1 year.
  Retrospective data collection from patient's medical records in mupirocin group Prospective data collection from patient's medical records in gentamicin group
Number and percentage Causative pathogens of Infectious peritonitis in mupirocin compared with gentamicin group | All pathogenic organisms of infectious peritonitis episodes occurred last year in mupirocin group and all pathogenic organisms of infectious peritonitis episodes have occurred after apply 0.1% grntamicin cream for 1 year.
  Retrospective data collection from patient's medical records in mupirocin group Prospective data collection from patient's medical records in gentamicin group
Percentage of catheter removal due to peritoneal dialysis-related infection | Retrospective period at least 1 year before recruit to the study, Prospective period at least 1 year after entry to the study.
  Prospective data collection from patient's medical records in gentamicin group
Time to first peritoneal dialysis-related infection after gentamicin application | Prospective period at least 1 year after entry to the study.
  Retrospective data collection from patient's medical records in mupirocin group Prospective data collection from patient's medical records in gentamicin group. Peritoneal-related infection diagnosis by physicians. Prospective data collection from patient's medical records in gentamicin group
Drug susceptibility of causative pathogens of peritoneal dialysis-related infection | Retrospective period at least 1 year before recruit to the study, Prospective period at least 1 year after entry to the study.
  Drug susceptibility test by broth micro-dilution and E-test. Retrospective data collection from patient's medical records in mupirocin group Prospective data collection from patient's medical records in gentamicin group

CONTACTS AND LOCATIONS:
Overall Officials: Ittaprach Yimsuk, PharmD, Study Chair — College of Pharmacy, Rangsit university; Pamila Tasanavipas, MD, Study Director — Phramongkutklao hospital and College of Medicine; Daraporn Rungprai, BCP, Study Director — Faculty of Pharmacy, Silpakorn University; Wichai Santimaleeworagun, BCP, Study Director — Faculty of Pharmacy, Silpakorn University; Kulthida Chaijumroen, B.N.S., Principal Investigator — Phramongkutklao hospital and College of Medicine
Locations (1):
- Phramongkutklao Hospital, Ratchathewi, Bangkok, Thailand